CLINICAL TRIAL: NCT03902145
Title: LULUN PROJECT II - Cohort Follow-up Study
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: The Mathile Institute for the Advancement of Human Nutrition (Other); Universidad San Francisco de Quito (Other); University of California, Davis (Other); RTI International (Other)
Responsible Party: Sponsor
Other Study IDs: 201704100
Record Dates: First submitted 2019-04-01; First posted 2019-04-03 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Stunting
Keywords: Complementary Feeding; Animal Source Foods; Bone Age; Stunting; Ecuador; Follow Up Cohort
MeSH Terms: conditions — Growth Disorders | interventions — Eggs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention Group: Children previously in the intervention group received one egg per day for 6 months beginning when the child was between 6-9 months of age.
  Interventions: Other: Egg
- Control Group

INTERVENTIONS:
Other: Egg — One egg per day for 6 months
  Groups: Intervention Group

SUMMARY:
Child stunting and micronutrient deficiencies are a major problem in developing countries, affecting millions of children.

Beginning at 6 months children need foods to complement nutrients received through breastfeeding; however, complementary feeding diets are well-documented to be inadequate in the developing world. Eggs, which are widely available and low-cost relative to other highly nutritious foods are underutilized and could potentially improve child growth and development. Prior to the Lulun Project RCT, no research had been conducted to evaluate their efficacy in improving micronutrient status. Lulun filled an important gap in the literature by examining, through a randomized controlled trial, the effect of egg consumption on biochemical markers of choline, vitamin B12, lipids, and amino acids in young children in a poor rural area of Ecuador. However, there is still scarce data on how early child complementary feeding interventions, such as the Lulun egg intervention, might impact child growth long-term.

This study will be designed as a follow-up cohort study to the Lulun Project RCT conducted in Cotopaxi Province from March-December 2015. The proposed follow-up study will investigate the potential long-term impacts of the egg intervention on child growth. Children and mother (caregiver) dyads with endline anthropometric measures from Lulun Project will be invited to participate in the follow-up study. Data will be collected on demographic, socioeconomic, and environmental information, morbidities, and child diet (including egg preparation and consumption), as well as child anthropometry (height, weight, head circumference). Additionally, the study will pilot test and compare radiographic measures of child bone maturity and organ size (kidney, liver, and spleen) using an app-based ultrasound. Investigators from Universidad de San Franscisco de Quito (USFQ), Washington University in St. Louis, and Mathile Institute will collaborate to conduct the study.

This project will also include a gender assessment component designed to ascertain how gender norms may affect prospects for successful scale up of smallholder poultry production. To this end, qualitative data will be collected from a small sample of participating mothers (caregivers) and key community stakeholders, in the form of in-depth interviews and/or focus groups.

DETAILED DESCRIPTION:
All mother (caregiver)-child dyads from the Lulun RCT will be contacted by mobile phone and invited to participate. A community meeting will first be held including community leaders and Lulun Project participants to present findings and explain the new follow-up study, Lulun Project II. This will give mothers (caregivers) the opportunity over at least a one week period to decide whether or not to participate and to discuss with family and friends. A field study team consisting of two individuals who participated in first trial and two students from Washington University will then contact mothers or caregivers and asked to come to various community sites used in the Lulun Project. Using processes and protocols from the original trial, mothers (caregivers) will first go through the informed consent and enrollment processes.

Eligibility criteria will include: 1) participant in the Lulun Project I; and 2) child healthy, without fever or severely malnourished. Mothers or primary caregivers of children will be given a written informed consent statement in Spanish to read and sign, indicating their consent and consent on behalf of their child. If the mothers/primary caregiver is less than 18 years of age, informed consent process will be sought from their parents or guardians. Participants with limited literacy will be offered the option to have the statement read to them. Caregivers will be invited to ask any questions about the nature of the study during this time.

For the gender analysis component of the study, a small number (10-20) of prospective mother (caregiver) participants, their partners, and key stakeholders will be contacted by phone by the Field Manager who will explain the nature and (qualitative) method of this part of the study. They will be invited to participate. Consent process for mothers, partners, and community stakeholders will occur after they agree to participate and just prior to interview or focus group.

ELIGIBILITY:
Inclusion Criteria:

* Participant in the Lulun Project I
* Child healthy, without fever or severely malnourished

Exclusion Criteria:

* Child not previously in the Lulun Project I
* Child has fever or is severely malnourished

Ages: 30 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Lulun Project II is a longitudinal follow-up study of the Lulun Project, which was conducted in Cotopaxi Province, Ecuador.
Sampling Method: Non-Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Height for Age Z-Score | One time point

SECONDARY OUTCOMES:
Bone Age Z Score | One time point
Weight for Age Z Score | One time point
Weight for Height Z Score | One time point
BMI Z-Score | One time point
Head Circumference for Age Z-Score | One time point

CONTACTS AND LOCATIONS:
Overall Officials: Lora Iannotti, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Universidad San Francisco de Quito, Quito, Pichincha, Ecuador

IPD SHARING:
Plan to Share IPD: No